CLINICAL TRIAL: NCT02729519
Title: Implantation of the Transcatheter Aortic Prosthesis SAPIEN 3 With or Without Prior Balloon Predilatation
Brief Title: TAVI Without Balloon Predilatation (of the Aortic Valve ) SAPIEN 3
Acronym: DIRECTAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL15_0392; 2015-A01823-46 (Other: ANSM)
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2024-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): standard procedure TAVI performed with systematic pre dilatation (With prior balloon dilatation)
  Interventions: Procedure: TAVI
- Groupe B (Experimental): standard procedure TAVI performed without pre dilatation (Without prior balloon dilatation)
  Interventions: Procedure: TAVI

INTERVENTIONS:
Procedure: TAVI — standard procedure TAVI performed with systematic pre dilatation (With prior balloon dilatation) (ARM A) ou without pre dilatation (ARM B)

SUMMARY:
Balloon predilatation of the aortic valve has been regarded as an essential step during the transcatheter aortic valve implantation (TAVI) procedure. However, recent evidence suggested that aortic valvuloplasty may be harmful and that high success rate may be obtained without prior dilatation of the valve. We hypothesize that TAVI performed without predilatation and using new generation balloon expandable prothesis is associated with a better net clinical benefit in comparison with procedure performed with pre dilatation.

DETAILED DESCRIPTION:
Background Transcatheter aortic valve implantation (TAVI) is now the standard of care for inoperable patients with severe symptomatic aortic stenosis and an accepted alternative to surgery for high-risk patients. Despite a high procedure success rate (> 95%), TAVI remained associated with complications directly related to the technique (stroke, aortic regurgitation, vascular access bleeding) or to co morbidities frequently associated with aortic valve disease in elderly and frail patients. Reducing periprocedural complications is thereby the key for the future use of TAVI in lower-risk patients.

Methods/design The transcatheter aortic valve implantation without prior balloon dilatation (DIRECTAVI) trial is a randomized controlled open label trial that include 240 patients randomized to TAVI performed with prior balloon dilatation of the valve (control arm) or direct implantation of the valve (test arm). The trial tests the hypothesis that the strategy of direct implantation of the balloon expandable SAPIEN 3 prosthesis is non-inferior to current medical practice using predilatation of the valve. The primary endpoint is related to immediate procedural success criteria and secondary end points include complications at 30-day follow-up (VARC 2 criteria). A subgroup analysis evaluates neurological ischemic events with cerebral MRI imaging (25 patients in each strategy group) performed before and after the procedure.

In conclusion, we hope that the study will provide robust evidence of safety and efficiency of TAVI performed without prior dilatation of the aortic valve using the balloon expandable SAPIEN 3 THV and will allow the interventional cardiologist to use this strategy in everyday practice.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Aortic valve stenosis with an aortic valve area <1 cm2 (<0,6 cm3/m2)
* Males or females of at least 18 years of age
* Logistic EuroSCORE ≥15% and/or a significant contraindication for open heart surgery (e.g., porcelain aorta or severe COPD) or all patients considered as having excessive surgical risk by the heart team
* Signed informed consent
* TAVI performed via transfemoral, sub clavicular or transaortic route with the SAPIEN 3 THV (Edwards Lifescience)

Exclusion Criteria:

* Transapical TAVI
* Preexisting aortic prosthesis (valve in valve technique)
* Vascular conditions that make insertion and endovascular access to the aortic valve impossible
* BAV performed for less than one week
* Recent myocardial infarction (STEMI within the last 3 months)
* Left ventricular or atrial thrombus by echocardiography
* Mitral or tricuspidal valvular insufficiency (> grade II)
* Evolutive or recent cerebrovascular event (within the last 3 months)
* Symptomatic carotid or vertebral arterial narrowing (>70%) disease
* Bleeding diathesis or coagulopathy or patient refusing blood transfusion
* Lack of written informed consent, severe mental disorder, drug/alcohol addiction
* Life expectancy < 1 year
* Hypersensitivity or contraindication to acetyl salicyl acid, heparin, ticlopidine, clopidogrel, or sensitivity to contrast media that cannot be adequately premedicated
* Participation in another drug or device study that would jeopardize the appropriate analysis of end-points of this study.
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
immediate procedural success | up to 72h
  Composite endpoint : absence of immediate procedural mortality AND correct positioning of a single prosthetic heart valve into the proper anatomical location AND intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient<20 mm Hg or peak velocity<3 m/s), AND no moderate or severe prosthetic valve regurgitation.

SECONDARY OUTCOMES:
cardiovascular event | 1 month
Complications post-procedure | up to 1 month
  VARC-2 criteria : life-threatening/major/minor bleeding, vascular access complications, heart failure, acute kidney failure (RANKIN classification stage 2 or 3), conduction disturbances, stroke, pacemaker implantation, Repeat procedure for valve-related dysfunction (surgical or interventional therapy)

OTHER OUTCOMES:
neurological ischemic events | up to 2 days
  Ancillary study : subgroup analysis evaluates neurological ischemic events with cerebral MRI imaging (25 patients in each strategy group) performed before and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Florence LECLERCQ, MD,PhD, Principal Investigator — UH of Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Robert P, Akodad M, Lattuca B, Gandet T, Meunier PA, Macia JC, Schmutz L, Steinecker M, Roubille F, Cayla G, Leclercq F. Balloon predilation or direct valve implantation in TAVI for women: Insights from the DIRECTAVI study. Catheter Cardiovasc Interv. 2024 Jul;104(1):97-104. doi: 10.1002/ccd.31086. Epub 2024 May 19. PMID 38764290
- [Derived] Jammoul N, Dupasquier V, Akodad M, Meunier PA, Moulis L, Soltani S, Macia JC, Robert P, Schmutz L, Steinecker M, Piot C, Targosz F, Benkemoun H, Lattuca B, Roubille F, Cayla G, Leclercq F. Long-term follow-up of balloon-expandable valves according to the implantation strategy: insight from the DIRECTAVI trial. Am Heart J. 2024 Apr;270:13-22. doi: 10.1016/j.ahj.2024.01.005. Epub 2024 Jan 20. PMID 38253304
- [Derived] Akodad M, Roubille F, Marin G, Lattuca B, Macia JC, Delseny D, Gandet T, Robert P, Schmutz L, Piot C, Maupas E, Robert G, Targosz F, Albat B, Cayla G, Leclercq F. Myocardial Injury After Balloon Predilatation Versus Direct Transcatheter Aortic Valve Replacement: Insights From the DIRECTAVI Trial. J Am Heart Assoc. 2020 Dec 15;9(24):e018405. doi: 10.1161/JAHA.120.018405. Epub 2020 Dec 10. PMID 33297821
- [Derived] Leclercq F, Robert P, Akodad M, Macia JC, Gandet T, Delseny D, Chettouh M, Schmutz L, Robert G, Levy G, Targosz F, Maupas E, Roubille F, Marin G, Nagot N, Albat B, Lattuca B, Cayla G. Prior Balloon Valvuloplasty Versus Direct Transcatheter Aortic Valve Replacement: Results From the DIRECTAVI Trial. JACC Cardiovasc Interv. 2020 Mar 9;13(5):594-602. doi: 10.1016/j.jcin.2019.12.006. PMID 32139216
- [Derived] Leclercq F, Robert P, Labour J, Lattuca B, Akodad M, Macia JC, Gervasoni R, Roubille F, Gandet T, Schmutz L, Nogue E, Nagot N, Albat B, Cayla G. Prior balloon valvuloplasty versus DIRECT transcatheter Aortic Valve Implantation (DIRECTAVI): study protocol for a randomized controlled trial. Trials. 2017 Jul 4;18(1):303. doi: 10.1186/s13063-017-2036-y. PMID 28676065